CLINICAL TRIAL: NCT00790374
Title: A Phase I Dose Escalating Study Evaluating the Pharmacodynamic Profile and Safety of BN83495 in Patients With Prostate Cancer With Evidence of Disease Progression While on Androgen Ablative Therapy
Brief Title: BN83495 in Prostate Cancer
Acronym: STX64PC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X-52-58064-003
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Pharmacodynamic profile and safety of BN83495
MeSH Terms: conditions — Prostatic Neoplasms | interventions — irosustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 6 patients have been enrolled, the cohort has been completed.
  Interventions: Drug: BN83495 (Cohort 1)
- Cohort 2 (Experimental): 6 patients have been enrolled in cohort 2, the cohort has been completed.
  Interventions: Drug: BN83495 (Cohort 2)
- Cohort 3 (Experimental): 5 patients have been enrolled in cohort 3. The cohort was closed after the 5th patient enrolled.
  Interventions: Drug: BN83495 (Cohort 3)

INTERVENTIONS:
Drug: BN83495 (Cohort 1) — 20 mg daily BN83495 for 28 days
  Arms: Cohort 1
Drug: BN83495 (Cohort 2) — 40 mg daily BN83495 for 28 days
  Arms: Cohort 2
Drug: BN83495 (Cohort 3) — 60 mg daily BN83495 for 28 days
  Arms: Cohort 3

SUMMARY:
The purpose of the study is to evaluate the pharmacodynamic profile and safety of BN83495 in patients with prostate cancer with disease progression while on androgen ablative therapy

DETAILED DESCRIPTION:
Evaluate the PD profile of BN83495 after 28 days of daily oral administration in patients with locally advanced or metastatic prostate cancer on androgen ablative therapy and with rising prostatic specific antigen

ELIGIBILITY:
Inclusion Criteria:

* Confirmed and locally advanced or metastatic prostate cancer with rising prostate-specific antigen (PSA), while on androgen ablative therapy.
* Over age 18.
* Demonstrated PSA "biochemical failure".
* Adequate bone marrow and hepatic function

Exclusion Criteria:

* Luteinizing Hormone-Releasing Hormone analogue treatment and treated with more than one additional second line of endocrine therapy
* Prior treatment with ketoconazole
* Prior chemotherapy for hormone refractory prostate cancer
* Pre-existing cardiac failure and/or clinically significant abnormal ECG or Echo

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Absolute and percentage change in levels of hormones from baseline to D28/29 at 6 timepoints | 28 days

SECONDARY OUTCOMES:
Tolerance (Physical Exam, ECOG Performance Status, Electrocardiogram, biochemistry/haematology, Urinalysis, Adverse Events, Concomitant Medications, disease progression) | Each visit through day 28/29
Pharmacokinetic assessments/Pharmacodynamic assessments | Pre-determined timepoints from baseline to day 28/29

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- United States (3):
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Duke University Medical Center United States, Durham, North Carolina
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin